CLINICAL TRIAL: NCT07027501
Title: The Evaluation of the Effectiveness of Febrile Seizure Training Given to Parents of Children Aged 6 Months to 5 Years
Brief Title: The Evaluation of the Effectiveness of Febrile Seizure Training Given to Parents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, TUĞÇE ŞİRİN, Principal Investigator, Zonguldak Bulent Ecevit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZBEU-TUGCE SIRIN-001; ZBEU (Other: ZONGULDAK BULENT ECEVIT UNIVERSITY)
Record Dates: First submitted 2025-05-21; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Febrile Convulsion
Keywords: febrile convulsion, fever, education, QR
MeSH Terms: conditions — Seizures, Febrile; Fever

STUDY DESIGN:
Intervention Model Description: The study included two groups: an intervention group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control (Other): No video-based educational intervention was administered to the control group
  Interventions: Other: The video based education group

INTERVENTIONS:
Other: The video based education group — The parents in the intervention group were provided with a video-based educational material on febrile seizures, which they accessed via a QR code.

SUMMARY:
Objective: The aim of this study was to evaluate the effectiveness of a video-based educational intervention delivered via QR code to parents of hospitalized children aged 6 months to 5 years-an age group in which febrile seizures are most commonly observed.

DETAILED DESCRIPTION:
Method: This study will be designed as a randomized controlled trial. The study population will consist of parents of children aged between 6 months and 5 years who are hospitalized in the pediatric wards of Kdz. Eregli State Hospital during the data collection period (September 1, 2024 - September 1, 2025). The sample will include 100 parents-50 in the intervention group and 50 in the control group-who meet the inclusion criteria.

Eligibility criteria for sampling; The child must have been hospitalized. The child must be between 6 months and 5 years of age. The parent must be able to speak and understand Turkish. The parent must agree to participate in the study Data collection: Between September 1, 2024, and September 1, 2025, the "Child and Parent Introductory Information Form" and the "Febrile Convulsion Knowledge Level Scale for Parents/Caregivers" will be completed by participants who meet the eligibility criteria.

No educational session or brochure will be provided to the control group. In the intervention group, after completing the "Child and Parent Introductory Information Form " and the "Febrile Convulsion Knowledge Level Scale for Parents/Caregivers", participants will be shown the educational brochure and granted access to the video training via the QR code included in the brochure.

At the end of the training, the "Febrile Convulsion Knowledge Level Scale for Parents/Caregivers" will be administered again. The brochure used in the training will be distributed to all participants in the intervention group.

Four weeks after the training, participants in the intervention group will be contacted again, and their data will be recollected using the same scale to assess knowledge retention and the long-term effectiveness of the training. Similarly, in the control group, the "Febrile Convulsion Knowledge Level Scale for Parents/Caregivers "will be re-administered four weeks after the initial data collection.

Data Analysis:

The data will be analyzed using the SPSS version 27.0 software.

ELIGIBILITY:
Inclusion Criteria:

The child has been hospitalized. The child is between 6 months and 5 years old. The parent can speak and understand Turkish. The parent agrees to participate in the study.

Exclusion Criteria:

The child has not been hospitalized. The child is younger than 6 months. The child is older than 5 years. The parent or legal guardian cannot speak or understand Turkish. The parent does not agree to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure Title: Change in Knowledge Levels Regarding Febrile Seizures Among Parents, Measured by the Febrile Seizure Knowledge Assessment Questionnaire | Knowledge scores were measured at baseline, immediately after training (1 hour later), and 4 weeks later in both intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data collected include sensitive personal and health information, and participants were not explicitly informed or consented to data sharing beyond the scope of this study. Therefore, to protect participant confidentiality and comply with ethical guidelines, the IPD will not be shared with other researchers.